CLINICAL TRIAL: NCT03085992
Title: Open-label Phase II Study of Induction Treatment With Folfoxiri Plus Bevacizumab Followed by Preoperative Chemoradiotherapy Plus Bevacizumab in Patients With Locally Advanced, Resectable Rectal Cancer.
Brief Title: Folfoxiri Plus Bevacizumab Followed by Chemoradiotherapy Plus Bevacizumab in Patients With Resectable Rectal Cancer
Acronym: TRUST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Alfredo Falcone, Prof., Azienda Ospedaliero, Universitaria Pisana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRUST; 2011-003340-45 (EudraCT Number)
Record Dates: First submitted 2016-06-08; First posted 2017-03-22 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; FOLFOXIRI; bevacizumab; trust
MeSH Terms: conditions — Rectal Neoplasms | interventions — Bevacizumab; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): INDUCTION TREATMENT WITH FOLFOXIRI PLUS BEVACIZUMAB FOLLOWED BY PREOPERATIVE CHEMORADIOTHERAPY PLUS BEVACIZUMAB
  Interventions: Drug: FOLFOXIRI plus Bevacizumab; Other: Chemoradiotherapy plus Bevacizumab

INTERVENTIONS:
Drug: FOLFOXIRI plus Bevacizumab — * BEVACIZUMAB 5 mg/kg over 30 minutes, day 1
  * IRINOTECAN 165 mg/sqm IV over 1-h, day 1
  * OXALIPLATIN 85 mg/sqm IV over 2-h, day 1
  * L-LEUCOVORIN 200 mg/sqm IV over 2-h, day 1
  * 5-FLUOROURACIL 3200 mg/sqm IV 48-h continuous infusion, starting on day 1 administered every two weeks for 6 cycles (3 months).
Other: Chemoradiotherapy plus Bevacizumab — * FLUOROURACIL 225 mg/sqm/day by protracted IV continuous infusion or -CAPECITABINE 825 mg/sqm/bid p.o. continuously without interruption for all the duration of radiation treatment;
  * EXTERNAL-BEAM IRRADIATION 50.4 GY in 28 daily fractions over 5.5 weeks;
  * BEVACIZUMAB 5 mg/kg over 30 minutes, starting on day 1 of radiation treatment day 1 and then every two weeks (for 3 cycles).

SUMMARY:
This study includes patients affected by advanced and resectable rectal adenocarcinoma. It provides an induction chemotherapy with FOLFOXIRI regimen plus Bevacizumab followed by Chemoradiotherapy plus Bevacizumab. Surgery with total mesorectal incision must be performed within 7-9 weeks after this last treatment. The protocol will be evaluate the disease free survival at two years. Translational analyses will be performed to show the presence of VEGF polymorphism, CD133 surface markers on colorectal CSCs.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of rectal adenocarcinoma. Diagnosis obtained by a biopsy technique which leaves the major portion of the tumor intact.
* Locally advanced, resectable disease defined by the presence of at least one of the following features: tumour extending to within 1 mm of or beyond the mesorectal fascia (ie, circumferential radial margin threatened or involved); lower third (≤ 6 cm from the anal verge) cT3 tumours; tumour extending 5 mm or more into perirectal fat; T4 tumour (ie, invading surrounding structures or peritoneum); clinical stage III disease (T1-4, N1-2), with the definition of a clinically positive lymph node being any node ≥ 1.0 cm;
* Distal border of the tumor must be located < 12 cm from the anal verge.
* No evidence of metastatic disease by CT scan of the chest and abdomen and total body PET-CT scan.
* Tumor must be amenable to curative resection (curative resection can include pelvic exenteration).
* No history of invasive rectal malignancy, regardless of disease-free interval.
* No other rectal cancers (i.e., sarcoma, lymphoma, carcinoid, squamous cell carcinoma, or cloacogenic carcinoma) or synchronous colon cancer.
* No clear indication of involvement of the pelvic side walls by imaging.
* Age between 18 and 75 years.
* ECOG Performance status < 2 if age < 70 years and = 0 if age 71-75 years.
* Life expectancy of at least 5 years (excluding diagnosis of cancer).
* Hematopoietic: absolute neutrophil count ≥ 1,000/mm3; platelet count ≥ 100,000/mm3; haemoglobin level ≥ 10 g/dL.
* Hepatic: total bilirubin ≤ 1.5 times upper limit of normal (ULN); alkaline phosphatase ≤ 2 times ULN; AST ≤ 2 times ULN. [Note: *If AST>ULN, serologic testing for Hepatitis B and C must be negative].
* Renal: creatinine clearance > 50 mL/min; no renal disease that would preclude study treatment or follow-up.
* Written informed consent to experimental treatment and pharmacogenomic analyses.

Exclusion Criteria:

* Previous treatment with oxaliplatin, irinotecan or bevacizumab. Previous 5-fluorouracil or capecitabine treatment is allowed.
* Previous pelvic radiation therapy.
* Hepatic disease that would preclude study treatment or follow-up; uncontrolled coagulopathy; history of viral hepatitis or other chronic liver disease.
* Cardiovascular disease that would preclude study treatment or follow-up; New York Heart Association class III or IV heart disease; active ischemic heart disease; myocardial infarction within the past 6 months; symptomatic arrhythmia; uncontrolled hypertension.
* Lack of upper gastrointestinal tract integrity or malabsorption syndrome; active inflammatory bowel disease (i.e., patients requiring current medical interventions or who are symptomatic).
* Pregnant or lactating women. Fertile patients must use effective contraception (i.e double-barrier contraceptive measures, oral contraception or avoidance of intercourse during the study and for 30 days after surgery).
* Patients with prior malignancies (with the exception of rectal cancer), including invasive colon cancer, are eligible provided they have been disease-free for ≥ 5 years and are deemed by their physician to be at low risk for recurrence.
* Other malignancy within the past 5 years with the exception of effectively treated squamous cell or basal cell skin cancer, melanoma in situ, carcinoma in situ of the cervix, or carcinoma in situ of the colon or rectum.
* Known hypersensitivity to fluorouracil, oxaliplatin or irinotecan or to Chinese hamster ovary cell proteins.
* Clinically significant peripheral neuropathy (i.e., neurosensory or neuromotor toxicity ≥ grade 2).
* Psychiatric or addictive disorders, or other conditions that, in the opinion of the investigator, would preclude study participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-03; Primary Completion 2017-07 (Actual); Study Completion 2018-03-12 (Actual)

PRIMARY OUTCOMES:
Disease-free survival rate at 2 years | Up to 2 years
  Disease-free survival is defined as time from study entry until progression of disease (according to RECIST 1.1) or death from any cause. Patients who are alive without having progressed at the end of the study will be censored at their last radiological assessment.

SECONDARY OUTCOMES:
Response rate | Up to 2 years
  Response rate is defined as the fraction of treated patients who achieve a response as defined according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria vers. 1.1.
Toxicity Rate | Up to 2 years
  Toxicity Rate is defined as the percentage of patients, relative to the total of enrolled subjects, experiencing treatment-related adverse events as assessed by National Cancer Institute Common Toxicity Criteria (version 3.0), during induction and concomitant chemoradiotherapy
Overall survival | Up to 2 years
  Overall survival is defined as the time from study entry until death from any cause. Patients who are alive at the end of the study will be censored at that point.
Pathological complete response rate | Up to 2 years
  Pathological complete response rate is defined as the fraction of treated patients who achieve pathological response after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Falcone, MD, Principal Investigator — Polo Oncologico Area Vasta Nord Ovest
Locations (4):
- Italy (4):
  - Irccs Istituto Oncologico Veneto, Padua
  - Polo Oncologico Area Vasta Nord Ovest, Pisa
  - ausl5 di Pisa, Pontedera
  - Dipartimento Oncologico AUSL 7, Siena

IPD SHARING:
Plan to Share IPD: Undecided